CLINICAL TRIAL: NCT00834600
Title: A Clinical Trial of Renin Profiling in Selection of Initial Antihypertensive Drug
Brief Title: Renin Profiling in Selection of Initial Antihypertensive Drug
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Louis & Rachel Rudin Foundation (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Michael H. Alderman, Professor of Epidemiology and Population Health, The Louis & Rachel Rudin Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-074; MMC #05-02-054
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — olmesartan; Hydrochlorothiazide; Amlodipine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCTZ , ARB (Experimental): Patients randomized to the Experimental Arm have initial drug choice determined by Plasma Renin Activity level. Low renin subjects are assigned to the diuretic hydrochlorothothiazide. Those with PRA >.65 ng/hr are assigned to the angiotensin receptor blocker, olmesartan.
  Interventions: Drug: olmesartan, hydrochlorothiazide, amlodipine; Drug: hydrochlorothiazide (HCTZ) or olmesartan
- Conventional antihypertensive therapy (Active Comparator): All patients randomized to Active Comparator Arm received hydrochlorothiazide 25 mg, which is increased to 50 mg at 3-4 weeks. At 6 weeks, olmesartan may be added if BP > 140 mmHg
  Interventions: Drug: olmesartan, hydrochlorothiazide, amlodipine; Drug: hydrochlorothiazide (HCTZ) or olmesartan

INTERVENTIONS:
Drug: olmesartan, hydrochlorothiazide, amlodipine — hydrochlorothiazide (HCTZ) 25mg OD, increased to 50 mg OD at 3 weeks. Olmesartan 20 mg OD, to be increased to 40 mg at 3 weeks. Amlodipine 5 mg, may be added at 6 weeks, if BP >140 mmHg
  Other Names: Renin guided selection of treatment
Drug: hydrochlorothiazide (HCTZ) or olmesartan — HCTZ 25 mg, increasing to 50 mg at 3-4 weeks or Olmesartan 20 mg, increasing to 40 mg at 3-4 weeks. If blood pressure >140/90 mmHg at 6 weeks, amlodipine 5 mg may be added
  Other Names: Standard Therapy

SUMMARY:
The purpose of this research study is to determine whether a simple blood test measuring a hormone called renin can better determine which first drug would be most effective in controlling blood pressure, in comparison with the more traditional approach recommended by JNC7 (Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure).

DETAILED DESCRIPTION:
Hypothesis: That antihypertensive drug selection guided by activity of the renin angiotensin system will be superior to the strategy advocated in JNC 7 in achieving blood pressure control on monotherapy.

Background: the National Heart, Lung, and Blood Institute, through the Joint National Committee on the Detection, Treatment and Control of Hypertension (JNC 7) has recommended that most hypertensive patients begin therapy with a diuretic and sequentially add other classes of drugs until blood pressure is controlled. This approach appears to assume homogeneity in the mechanism by which BP is controlled in different patients. When this standardized strategy has been rigidly applied in Clinical Trials, a majority of patients generally require 2 or more agents to achieve blood pressure control.

The pioneering work of Laragh, Sealey and their colleagues, widely confirmed by others, suggests instead that heterogeneity, in fact, characterizes patterns of blood pressure control in populations. This heterogeneity can be exposed through assessment of the activity of the renin angiotensin system (RAS). Specifically, volume and vasoconstriction determine blood pressure control. Patients in whom volume predominates have suppressed RAS, and, conversely, those in whom vasoconstriction predominates will have an activated RAS. This can be simply and accurately determined by estimation of plasma renin activity (PRA).

It has been demonstrated that volume and vasoconstriction dependent hypertensive patients respond best to different drugs. By exploitation of the RAS it is possible to provide rational therapy to each patients according to the mechanism by which blood pressure is controlled. The result is that appropriate therapy can be both more effective and more efficient. A specific system the Laragh Method has been designed to translate this physiologically based paradigm into a practical scheme or patient management.

The purpose of this trial is to determine whether the Laragh Method will lead to better and more efficient blood pressure control in a general population of hypertensive patients than does the existing treatment strategy. The measure by which this hypothesis will be tested is percentage of hypertensive patients achieving blood pressure control on monotherapy.

The significance of this trial is enormous for both individuals and society. Some 50 million Americans have hypertension and more than 25 million are currently in treatment. If the Laragh Method leads to more parsimonious and effective care, it will mean literally millions of individual patients will be spared the burden of unnecessary polypharmacy. Moreover, the strain on health care costs associated with antihypertensive therapy will be redu

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 40 to 85 years of age
* Sustained systolic blood pressure between 140-180 mm Hg
* Free of antihypertensive therapy at randomization for at least 4 weeks

Exclusion criteria:

* Ages <40, or >85 years
* Systolic blood pressure >180 mm Hg
* Blood pressure >180/105 mm Hg during the washout period
* Require antihypertensive agents for non-blood pressure indications
* Taking clonidine
* On a beta-blocker drug and have known or suspected coronary artery disease
* Documented history of a heart attack, new onset of chest pain, or a coronary revascularization procedure within the past year, congestive heart failure
* Serious intercurrent illness
* An active ulcer
* Have certain abnormal laboratory tests (elevated serum creatinine >1.5 mg/dl, transaminase > 2 times upper limit of normal or active liver disease),
* Hypersensitivity, allergy or have an intolerance to angiotensin II receptor blockers (olmesartan), hydrochlorothiazide or amlodipine
* Mentally or legally unable to participate
* Have or are currently abusing alcohol, have abused drugs within the past 2 years
* Have been in another drug study in the past month.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2005-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Percent of patients with BP <140/90 mmHg and on monotherapy at the 5th visit. | 3-4 months

SECONDARY OUTCOMES:
Will include change in blood pressure, percent of patients with blood pressure <140/mmHg, total number of classes of antihypertensive agents taken, adverse events and discontinuation of therapy. | 3-4 months
In addition, we will be able to determine the reproducibility of PRA determination in this clinical setting. Finally, it will be possible to demonstrate the value of "in-treatment" PRA as a guide to treatment modification. | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Alderman, M.D., Principal Investigator — Albert Einstein College of Medicine
Locations (5):
- United States (5):
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Albert Einstein College of Medicine - GCRC, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Bronx Nephrology Hypertension, PC, The Bronx, New York
  - Ralph Yung, MD, The Bronx, New York

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Laragh JH: Laragh's Lessons in Renin System Pathophysiology for Treating Hypertension and its Fatal Cardiovascular Consequences. Elsevier Science Inc.,2002,N.Y.
- [Background] Laragh JH, Sealey JE. Renin system understanding for analysis and treatment of hypertensive patients: a means to quantify the vasoconstrictor elements, diagnose curable renal and adrenal causes, assess risk of cardiovascular morbidity, and find the best-fit drug regimen. Chapter 107, In: Hypertension:Pathophysiology Diagnosis and Management, 2nd Edition, Edited by JH Laragh and BM Brunner. Raven Press,Ltd.,New York 1995.
- [Background] Sealey JE. Measurement of the hormones of the renin system in hypertensive patients. Clin Biochem. 1981 Oct;14(5):273-81. doi: 10.1016/s0009-9120(81)91000-6. No abstract available. PMID 6120769